CLINICAL TRIAL: NCT05758090
Title: Comparison of Newborn Infant Parasympathetic Evaluation (NIPE) Index Versus Standard Hemodynamic Response for Guiding Intraoperative Fentanyl Administration in Children Younger Than 2 Years Under General Anesthesia
Brief Title: Newborn Infant Parasympathetic Evaluation (NIPE) for Guiding Intraoperative Fentanyl in Children Under 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE651243
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain; Analgesia; Children, Only; Narcotic Use
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group NIPE (Experimental): Intraoperative fentanyl administration will be guided by NIPE protocol
  Interventions: Procedure: NIPE monitor
- Group Control (Placebo Comparator): Intraoperative fentanyl administration will be guided by clinical signs
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: NIPE monitor — Procedure/Surgery: NIPE protocol. Give intraoperative fentanyl according to NIPE value. NIPE score 50-70 indicates optimal narcotic effect. NIPE score > 70 indicated overdosage of narcotic and narcotic should be withheld. NIPE score < 50 indicates inadequate narcotic and narcotic should be given.
  Arms: Group NIPE
Procedure: Control — Procedure/Surgery: Standard protocol. Give intraoperative fentanyl according to vital signs.
  Arms: Group Control

SUMMARY:
During general anesthesia, objective monitoring for analgesia is still lacking. The administration of opioids relies on the experience of the anesthesiologist. There are some monitors, e.g., Analgesia Nociception Index (ANI), showing that they can evaluate analgesia in adults. Recently, a Newborn Infant Parasympathetic Evaluation (NIPE) monitor was released for assessing analgesia in children with age less than 2 years. The investigators aim to assess the efficacy of NIPE as a guide for intraoperative fentanyl administration in children under 2 years.

DETAILED DESCRIPTION:
During balanced anesthesia, hypnosis can be monitored with BIS, muscle relaxation can be monitored with a train-of-four, however, analgesia lacks precise monitoring. The anesthesiologist administers narcotics according to clinical signs and experience. Analgesia Nociception Index (ANI) has been introduced as an objective monitor for analgesia in adults. Recently, a Newborn Infant Parasympathetic Evaluation (NIPE) monitor has been introduced to assess analgesia in children under 2 years, however, clinical studies regarding its clinical efficacy are scarce.

The objective of this study is to assess the efficacy of NIPE as a guide for intraoperative fentanyl administration in children under 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newborn up to 2 years old
* ASA Status 1-2
* Undergoing elective surgery of upper part of body

Exclusion Criteria:

* Premature
* Arrhythmia
* Concomitant use of regional anesthesia
* Plan for ICU admission

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain: Face, Legs, Activity, Cry, Consolability scale (FLACC scale) | During 120 minutes in PACU
  Assess pain using a FLACC score every 15 minutes. FLACC has a range from 0 to 10 with 0 indicates no pain while 10 indicates worst pain. NRS of 0-3 is mild, 4-6 is moderate, and 7-10 is severe pain.

SECONDARY OUTCOMES:
Postoperative fentanyl consumption | During 120 minutes in PACU
  Fentanyl administration in PACU
Postoperative sedation score | During 120 minutes in PACU
  Sedation score (0-3; higher scores mean a worse outcome) in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, PhD, Study Chair — Khon Kaen University
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weber F, Roeleveld HG, Geerts NJE, Warmenhoven AT, Schroder R, de Leeuw TG. The heart rate variability-derived Newborn Infant Parasympathetic Evaluation (NIPE) Index in pediatric surgical patients from 0 to 2 years under sevoflurane anesthesia-A prospective observational pilot study. Paediatr Anaesth. 2019 Apr;29(4):377-384. doi: 10.1111/pan.13613. Epub 2019 Mar 21. PMID 30793426
- [Result] Recher M, Boukhris MR, Jeanne M, Storme L, Leteurtre S, Sabourdin N, De Jonckheere J. The newborn infant parasympathetic evaluation in pediatric and neonatology: a literature review. J Clin Monit Comput. 2021 Oct;35(5):959-966. doi: 10.1007/s10877-021-00670-8. Epub 2021 Feb 15. PMID 33590418
- [Result] Lim BG. Nociception monitoring tools using autonomic tone changes for intraoperative analgesic guidance in pediatric patients. Anesth Pain Med (Seoul). 2019 Oct 31;14(4):380-392. doi: 10.17085/apm.2019.14.4.380. PMID 33329766
- [Result] Zhang K, Wang S, Wu L, Song Y, Cai M, Zhang M, Zheng J. Newborn infant parasympathetic evaluation (NIPE) as a predictor of hemodynamic response in children younger than 2 years under general anesthesia: an observational pilot study. BMC Anesthesiol. 2019 Jun 11;19(1):98. doi: 10.1186/s12871-019-0774-y. PMID 31185928